CLINICAL TRIAL: NCT06986226
Title: MultiCPR: The Influence of Ventilations on Mental Arithmetics
Acronym: MultiCPR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mathias Maleczek, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: MultiCPR_2
Record Dates: First submitted 2025-04-29; First posted 2025-05-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Multitasking Behavior
MeSH Terms: conditions — Multitasking Behavior | interventions — Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilations/CPR (Active Comparator): Calculations made with/without performing ventilations - cross over design to decide what to do first, NASA-TLX will be measured
  Interventions: Behavioral: Dose Calculations; Procedure: Ventilations
- no ventilations/CPR (Active Comparator): Calculations made with/without performing ventilations - cross over design to decide what to do first, NASA-TLX will be measured
  Interventions: Behavioral: Dose Calculations

INTERVENTIONS:
Behavioral: Dose Calculations — Dose calculations either with or without performing ventilations during CPR (15:2)
Procedure: Ventilations — Performing ventilations during CPR in a 15:2 manner
  Arms: Ventilations/CPR

SUMMARY:
The purpose of this clinical study is to investigate how performing ventilations during pediatric resuscitation affects the ability to perform mental tasks. In particular, the effect on the participant's ability to perform dose calculations will be investigated. The aim is to draw conclusions about the effects of ventilations on other mental tasks.

How does the clinical trial work? This clinical trial will be conducted in several locations and will involve a total of 38 people. The study will be conducted by the Department of Anesthesiology of the Medical University of Vienna.

Participation in this clinical study is expected to last 30 minutes.

The following measures will be carried out exclusively for study reasons:

Depending on the sub-study you are participating in, different tasks will be performed:

Adult sub-study:

During this study, participants will be asked to perform mental arithmetic: Participants will be read a number every 2 seconds and have to add the last two in each case. The numbers are predetermined and randomly generated. At the end, we will evaluate how many results were correct.

ELIGIBILITY:
Inclusion:

* Healthy medical professionals trained in CPR (paramedics, prehospital emergency physicians, anesthesiologists, internal medicine doctors, nurses, midwifery students, pediatricians)
* CPR Training in the last four years
* Fit and rested.

Exclusion:

- Pregnant probands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-26 (Actual)

PRIMARY OUTCOMES:
Dose calculations | during 2x2 minutes of inclusion
  Number of correct calculations

SECONDARY OUTCOMES:
NASA-TLX | 4 minutes, 2 times in total per participant
  Nasa Task load index (min: 0, max: 120, higher scores mean higher cognitive load)

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Simulation Center, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No